CLINICAL TRIAL: NCT01512836
Title: A Randomized Controlled Trial to Determine Outcome and Cost Effectiveness of Case Management of Patients Suffering From Chronic Obstructive Pulmonary Disease (COPD) in a Danish Setting
Brief Title: A Randomized Controlled Trial to Determine Outcome and Cost Effectiveness of Case Management of Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kronikerenheden Nordjylland (Other Government)
Responsible Party: Principal Investigator, Sabrina Storgaard Soerensen, Ph.d. student, Kronikerenheden Nordjylland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RN-1
Record Dates: First submitted 2012-01-15; First posted 2012-01-19 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Case management; CEA; Health economy; Quality of Life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Case Management (Experimental): The patients who are randomized to the intervention group will be assigned to case management. The case manager is expected to integrate care from a health maintenance and promotion perspective, where the overall goal is the promote and support the patients self care (see intervention description).
  Interventions: Behavioral: Case Management
- Usual Care (No Intervention): Patients randomized to the usual care group will receive conventional health and social services. Patients in this group will not receive support from a case manager.

INTERVENTIONS:
Behavioral: Case Management — Patients, who are randomized to the intervention group, will receive case management from a trained and experienced nurse. The case manager will carry out following tasks:
  * Formulation and implementation of care plans together with the patient
  * Monitoring of individual status and care plan effectuation
  * Overall coordination between health care providers
  * Support to the patient and their caregivers during times of transition related to health status and environmental changes (e.g. hospital to home)
  * Regular telephone consultations and home visits
  * Promote disease-self management through coaching
  Other Names: Care management, integrated care, shared care
  Arms: Case Management

SUMMARY:
This randomized controlled trial (RCT) will examine a nurse case management model for patients suffering from chronic obstructive pulmonary disease (COPD) in a Danish municipality, and is performed in order to evaluate the use of case management as a tool in achieving integrated, quality and cost-effective care for this group of patients.

The main objectives are to evaluate how case management influences on hospital admissions, mortality, quality of life and self care, as well as to compare costs and cost-effectiveness of case management vs. usual care.

DETAILED DESCRIPTION:
Case management is being implemented as a health service strategy that should contribute to maximize health outcomes within a cost-constrained environment. Evaluations of case management in Danish settings are sparse, and so far no Danish studies have evaluated the cost-effectiveness of case management.

This study is performed as a RCT, and the study focuses exclusively on patients with COPD. The patients will be enrolled and randomized after being referred to rehabilitation at the local rehabilitation center in Aalborg municipality, Denmark. 150 patients will be randomly assigned to two groups of 75 patients each. Participants in the control group will receive usual care, whereas patients assigned to the interventional group will receive case management besides their usual care. Each patient will be followed for 12 months. Patients in both groups will fill out questionnaires at baseline and 12 months. The data register system "Health - Planning and Quality" in the Northern Region of Jutland will be used to determine health care services and costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are clinically referred to rehabilitation at Aalborg Rehabilitation Center for their diagnosed COPD

Exclusion Criteria:

* Patients living outside Aalborg municipality, or who is considering to move to another municipality or country in near future.
* Patients without a telephone
* Patients with dementia
* Patients participating in other research studies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
COPD hospitalization rates | 1 year (study inclusion - 12 months of follow-up)

SECONDARY OUTCOMES:
Mortality | 1 year (study inclusion - 12 months of follow-up)
Self Care | A baseline measure at study inclusion and after 12 months of follow-up
  The Patient-Activation Measure short form (PAM-13) will be used to evaluate change in self care. The investigators will obtain 2 measurements from each patient during the study period.
Quality of Life (QoL) | A baseline measure at study inclusion and after 12 months of follow-up
  The investigators will obtain 2 measurements from each patient and are therefore able to evaluate the change in Qol from baseline to end of study (1 year in total). Both generic (EQ-5D, SF-12) and disease-specific questionnaires (Sct. George Respiratory questionnaire, SG-RQ) will be used.
Cost-effectiveness of case management | 1 year
  The cost-effectiveness analysis will examine and compare the cost of health care resources and health outcomes between the two groups. The costs will include all health care utilization during the 1 year of follow-up.
  Quality adjusted life years (QALYs) is the preferred measure for cost-effectivenes analysis. QALYs will be calculated based on the EuroQol (EQ-5D).

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina S Sørensen, Ph.d., Principal Investigator — Kronikerenheden Nordjylland
Locations (1):
- Kronikerenheden, Nordjylland, Aalborg, Denmark

REFERENCES:
- [Derived] Sorensen SS, Pedersen KM, Weinreich UM, Ehlers L. Economic Evaluation of Community-Based Case Management of Patients Suffering From Chronic Obstructive Pulmonary Disease. Appl Health Econ Health Policy. 2017 Jun;15(3):413-424. doi: 10.1007/s40258-016-0298-2. PMID 27928660